CLINICAL TRIAL: NCT06828068
Title: Using Radiation-free Ultrasound for Screening Scoliosis Among Female School Children in Hong Kong to Reduce Unnecessary X-ray Exposure
Acronym: SScoE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Tsz-ping Lam, Associate Professor (Clinical) of Orthopaedics and Traumatology, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SScoE_Protocol_V01; Project no: 04152896 (Other Grant/Funding Number: Health and Medical Research Fund of the Hong Kong S.A.R., China)
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Scoliosis; Spinal Curvatures; Spinal Diseases; Bone Diseases; Musculoskeletal Disease
Keywords: Scoliosis, Ultrasound, screening program, immature female
MeSH Terms: conditions — Scoliosis; Spinal Curvatures; Spinal Diseases; Bone Diseases; Musculoskeletal Diseases | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SScoE (Other): This is a cross-sectional study on female screened school children recommended for radiographic assessment in the scoliosis screening program of SHS in Hong Kong. Both x-ray, ultrasound and ATR measurement of the spine will be performed on the same day at Prince of Wales Hospital.
  Interventions: Device: Ultrasound (Scolioscan system), and EOS radiography system

INTERVENTIONS:
Device: Ultrasound (Scolioscan system), and EOS radiography system — Scolioscan ultrasound system was reported to be reliable and valid for spinal deformity assessment. The system composes of an ultrasound scanner with a linear probe of 10 cm width and frequency range of 4-10MHz, a frame structure and a spatial sensor attached to the ultrasound probe for spatial data capture. Daily calibration will be performed using phantom to assure accuracy of spine image formation and subsequent angle measurement. Subjects will stand on the Scolioscan platform with a standardized posture kept stable with pegs throughout the scanning process. The probe will be steered from L5 to C7 spinous process for scanning. SPA will be used to determine the ultrasound-based Referral Status through predicting whether the Cobb angle is beyond the referral threshold of ≥20° or not. There are two values for the Referral Status: either "for specialist referral" or "not for specialist referral". Coronal Cobb angle measurement on EOS radiographs will be used as gold standard.

SUMMARY:
In the scoliosis screening program of the Student Health Service (SHS), Department of Health (DH), in Hong Kong, more than 50% of screened school children prescribed with x-ray examination basing on the screening protocol did not have Cobb angle greater than the referral threshold of 20°; ie they did not need specialist referral and thus were subjected to unnecessary x-ray exposure. Our primary objective is to determine whether a new radiation-free ultrasound system could identify subjects with Cobb angle greater than the referral threshold of 20° thus avoiding unnecessary x-rays in the referral workflow. The secondary objective is to evaluate if Angle of Trunk Rotation (ATR) can further increase the accuracy of ultrasound assessment.

This study is an extension of the registered project entitled "Using Radiation-free Ultrasound for Screening Scoliosis Among School Children in Hong Kong to Reduce Unnecessary X-ray Exposure", (ClinicalTrials.gov Identifier: NCT03135665), however focusing on validity of ultrasound measurement for immature female subjects aged around ten with year since menarche equal to or less than 9 months, who are prone to curve progression, and thus are among the most critical group in clinical management of scoliosis for regular monitoring, treatment decision, and brace indication.

ELIGIBILITY:
Inclusion Criteria:

i. School children in Hong Kong attending School Screening Program provided by Student Health Service ii. Recommended for radiographic assessment in the scoliosis screening program iii. Female with year since menarche of equal to or less than 9 months

Exclusion Criteria:

i. Patients with standing height <1 m, or >2 m ii. Patients with body mass index (BMI) ≥25 kg/m2 iii. Subjects with skin diseases iv. Subjects with fracture or wound that affect ultrasound scanning v. Subjects with ferromagnetic implants vi. Subjects with surgery done for the spine vii. Subjects with winged scapula or other irregularity of back contour that affect ultrasound scanning viii. Subjects who cannot stand steadily during scanning ix. Subjects with allergy to ultrasound gel

Ages: 8 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Female with year since menarche (YSM) of equal to or less than 9 months
Enrollment: 442 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ultrasound-based Referral Status | Baseline
  "for specialist referral" or "not for specialist referral", through predicting whether the Cobb angle is beyond the referral threshold of ≥20° or not in scoliosis screening

SECONDARY OUTCOMES:
Angle of Trunk Rotation (ATR) | Baseline
  evaluate if this parameter can increase the accuracy of ultrasound assessment

CONTACTS AND LOCATIONS:
Overall Officials: Tsz-ping Lam, FHKAM(Ortho Surg), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. COBB JR. The problem of the primary curve. J Bone Joint Surg Am. 1960 Dec; 42-A:1413-25. 2. Weinstein SL, Dolan LA, Wright JG, Dobbs MB. Effects of bracing in adolescents with idiopathic scoliosis. N Engl J Med. 2013 Oct 17; 369(16):1512-21. 3. Hresko MT, Talwalkar V, Schwend R; AAOS, SRS, and POSNA. Early Detection of Idiopathic Scoliosis in Adolescents. J Bone Joint Surg Am. 2016 Aug 17;98(16):e67. 4. Luk KD, Lee CF, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Fong DY. Clinical effectiveness of school screening for adolescent idiopathic scoliosis: a large population-based retrospective cohort study. Spine (Phila Pa 1976). 2010 Aug 1;35(17):1607-14. 5. Fong DY, Lee CF, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Luk KD. A meta-analysis of the clinical effectiveness of school scoliosis screening. Spine (Phila Pa 1976). 2010 May 1;35(10):1061-71. 6. Lee CF, Fong DY, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Luk KD. Costs of school scoliosis screening: a large, population-based study. Spine (Phila Pa 1976). 2010 Dec 15;35(26):2266-72. 7. Lee CF, Fong DY, Cheung KM, Cheng JC, Ng BK, Lam TP, Mak KH, Yip PS, Luk KD. Referral criteria for school scoliosis screening: assessment and recommendations based on a large longitudinally followed cohort. Spine (Phila Pa 1976). 2010 Dec 1;35(25):E1492-8. 8. Fong DY, Cheung KM, Wong YW, Wan YY, Lee CF, Lam TP, Cheng JC, Ng BK, Luk KD. A population-based cohort study of 394,401 children followed for 10 years exhibits sustained effectiveness of scoliosis screening. Spine J. 2015 May 1;15(5):825-33. 9. Hoffman DA, Lonstein JE, Morin MM, Visscher W, Harris BS 3rd, Boice JD Jr. Breast cancer in women with scoliosis exposed to multiple diagnostic x rays. J Natl Cancer Inst. 1989 Sep 6;81(17):1307-12. 10. Doody MM, Lonstein JE, Stovall M, Hacker DG, Luckyanov N, Land CE. Breast cancer mortality after diagnostic radiography: findings from the U.S. Scoliosis Cohort Study. Spine (Phila Pa 1976). 2000 Aug 15;25(16):2052-63. 11. Schmitz-Feuerhake I, Pflugbeil S. 'Lifestyle' and cancer rates in former East and West Germany: the possible contribution of diagnostic radiation exposures. Radiat Prot Dosimetry. 2011 Sep;147(1-2):310-3. doi: 10.1093/rpd/ncr348. Epub 2011 Aug 10. 12. Suzuki S, Yamamuro T, Shikata J, Shimizu K, Iida H. Ultrasound measurement of vertebral rotation in idiopathic scoliosis. J Bone Joint Surg Br. 1989 Mar;71(2):252-5. 13. Huang QH, Zheng YP, Lu MH, Chi ZR. Development of a portable 3D ultrasound imaging system for musculoskeletal tissues. Ultrasonics. 2005 Jan;43(3):153-63. 14. Cheung CW, Law SY, Zheng YP. Development of 3-D ultrasound system for assessment of adolescent idiopathic scoliosis (AIS): and system validation. Conf Proc IEEE Eng Med Biol Soc. 2013;2013:6474-7. doi: 10.1109/EMBC.2013.6611037. 15. Purnama KE, Wilkinson MH, Veldhuizen AG, van Ooijen PM, Lubbers J, Burgerhof JG, Sardjono TA, Verkerke GJ. A framework for human spine imaging using a freehand 3D ultrasound system. Technol Health Care. 2010;18(1):1-17. 16. Li M, Cheng J, Ying M, Ng B, Zheng YP, Lam TP, Wong WY, Wong MS. Could clinical ultrasound improve the fitting of spinal orthosis for the patients with AIS? Eur Spine J. 2012 Oct;21(10):1926-35. 17. Chen W, Lou EH, Zhang PQ, Le LH, Hill D. Reliability of assessing the coronal curvature of children with scoliosis by using ultrasound images. J Child Orthop. 2013 Dec;7(6):521-9. doi: 10.1007/s11832-013-0539-y. Epub 2013 Oct 22. 18. Ungi T, King F, Kempston M, Keri Z, Lasso A, Mousavi P, Rudan J, Borschneck DP, Fichtinger G. Spinal curvature measurement by tracked ultrasound snapshots. Ultrasound Med Biol. 2014 Feb;40(2):447-54. 19. Li M, Cheng J, Ying M, Ng B, Lam TP, Wong MS. A Preliminary Study of Estimation of Cobb's Angle From the Spinous Process Angle Using a Clinical Ultrasound Method. Spine Deform. 2015 Sep;3(5):476-482. 20. Cheung CW, Zhou GQ, Law SY, Mak TM, Lai KL, Zheng YP. Ultrasound Volume Projection Imaging for Assessment of Scoliosis. IEEE Trans Med Imaging. 2015 Aug;34(8):1760-8. 21. Zheng YP, Lee TT, Lai KK, Yip BH, Zhou GQ, Jiang WW, Cheung JC, Wong MS, Ng BK, Cheng JC, Lam TP. A reliability and validity study for Scolioscan: a radiation-free scoliosis assessment system using 3D ultrasound imaging. Scoliosis Spinal Disord. 2016 May 31;11:13. 22. Morrison DG, Chan A, Hill D, Parent EC, Lou EH. Correlation between Cobb angle, spinous process angle (SPA) and apical vertebrae rotation (AVR) on posteroanterior radiographs in adolescent idiopathic scoliosis (AIS). Eur Spine J. 2015 Feb;24(2):306-12. 23. Lowe T, Berven SH, Schwab FJ, Bridwell KH. The SRS classification for adult spinal deformity: building on the King/Moe and Lenke classification systems. Spine (Phila Pa 1976). 2006 Sep 1;31(19 Suppl):S119-25.